CLINICAL TRIAL: NCT00808483
Title: Effect of a Walking Skill Training Program in Patients Who Have Undergone Total Hip Arthroplasty: Followup One Year After Surgery
Brief Title: Walking Skill Training Program Effects in Patients With Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Kristi E Heiberg, PhD, Registrered physiotherapist, PhD, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008/2325
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Arthroplasty, Replacement, Hip; Exercise Therapy
Keywords: total hip arthroplasty; physical functioning; training program; self-efficacy; exercise therapy; walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Walking skill training group (Experimental): Participation in the supervised walking skill training program.
  Interventions: Other: Walking skill training program
- Control group (No Intervention): No participation in the supervised walking skill training program

INTERVENTIONS:
Other: Walking skill training program — 12 individualized training sessions containing functional exercises like walking, stair climbing, balance training and with supervision and guidance from a physiotherapist.
  Arms: Walking skill training group

SUMMARY:
Rehabilitation plays an important part after total hip arthroplasty. In this common practice few studies have been performed on this issue.

The aims of this study were:

1. to examine the immediate effects of a walking skill training program on walking, stair climbing, balance, self-reported physical functioning physical functioning, pain and self-efficacy compared to a control group without supervised physiotherapy
2. to examine whether the effects persisted 12 months after surgery

ELIGIBILITY:
Inclusion Criteria:

* Primary cox arthrosis
* Good written and oral Norwegian language

Exclusion Criteria:

* Severe hip arthrosis in the other hip or severe gon arthrosis that restricted walking
* Neurological disorders
* Rheumatoid arthritis

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristi E Heiberg, PhD, Principal Investigator — University of Oslo; Kristi E Heiberg, PhD, Principal Investigator — Bærum Hospital Vestre Viken
Locations (1):
- Department of health science, University of Oslo, Oslo, Oslo 0317, Norway

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the hospital the day before surgery from October 2008 to March 2010.
Groups:
- Walking Skill Training Group: 12 sessions of participation in the walking skill training program.
  Walking skill training program: 12 individualized training sessions containing functional exercises like walking, stair climbing, balance training and with guidance from a physiotherapist.
- Control Group: No participation in the walking skill training group
Period: From 3 to 5 Months After Surgery
Arm/Group | Walking Skill Training Group | Control Group
Started | 35 | 33
Completed | 33 | 32
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Period: From 5 Months to 12 Months
Arm/Group | Walking Skill Training Group | Control Group
Started | 33 | 32
Completed | 32 | 32
Not Completed | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Walking Skill Training Group: 12 sessions of participation in the walking skill training program.
  Walking skill training program: 12 individualized training sessions containing functional exercises like walking, stair climbing, balance training and sit-to-stand with guidance and supervision from a physiotherapist.
- Total: Total of all reporting groups
Arm/Group | Walking Skill Training Group | Control Group | Total
Number analyzed (Participants) | 35 | 33 | 68
Age, Continuous [Mean (Full Range); unit: years] | 65 [49 to 78] | 66 [45 to 81] | 66 [45 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 14 | 35
  Male | 14 | 19 | 33
BMI [Mean (Full Range); unit: kg/m^2] | 27 [20 to 37] | 27 [21 to 36] | 27 [20 to 37]

OUTCOME MEASURES:

1. Primary Outcome: 6 Minutes Walk Test (6MWT)
Description: Participants walked in a 40 meter hospital corridor for 6 minutes.
Time Frame: 5 months and 12 months
Measure: Mean (95% Confidence Interval); unit: meters
Groups:
- Walking Skill Training Group: 12 sessions of participation in the supervised walking skill training program.
  Walking skill training program: 12 individualized training sessions containing functional exercises like walking, stair climbing, balance training and with guidance from a physiotherapist.
- Control Group: No participation in the walking skill training program
Arm/Group | Walking Skill Training Group | Control Group
Number analyzed (Participants) | 35 | 33
meters
  6MWT at 5 months | 513 [497 to 529] | 462 [445 to 478]
  6MWT at 12 months | 535 [516 to 555] | 483 [463 to 503]

2. Secondary Outcome: Hip Dysfunction and Osteoarthritis Outcome Score (HOOS)
Description: Self-reported symptoms, pain, physical function, function in sport and recreation, quality of life. 0 (worse) - 100 (best)
Time Frame: 5 months and 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Walking Skill Training Group: 12 session of participation in the supervised walking skill training program
Arm/Group | Walking Skill Training Group | Control Group
Number analyzed (Participants) | 35 | 33
units on a scale
  HOOS pain at 5 months | 92 [89 to 95] | 90 [87 to 93]
  HOOS pain at 12 months | 94 [91 to 96] | 94 [92 to 97]

3. Secondary Outcome: Harris Hip Score (HHS)
Description: Pain and physical function. 0 (worse) - 100 (best)
Time Frame: 5 months and 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Walking Skill Training Group: 12 sessions of participation in a supervised walking skill training program
Arm/Group | Walking Skill Training Group | Control Group
Number analyzed (Participants) | 35 | 33
units on a scale
  HHS at 5 months | 93 [91 to 96] | 90 [87 to 92]
  HHS at 12 months | 96 [93 to 98] | 92 [90 to 95]

4. Secondary Outcome: Self-efficacy
Description: Self-reported self-efficacy in activities. 0 (worse) - 100 (best).
Time Frame: 5 months and 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Walking Skill Training Group: 12 sessions of participation in the supervised walking skill training group
Arm/Group | Walking Skill Training Group | Control Group
Number analyzed (Participants) | 35 | 33
units on a scale
  Self-efficacy at 5 months | 86 [82 to 90] | 81 [77 to 84]
  Self-efficacy at 12 months | 88 [83 to 92] | 84 [79 to 88]

5. Secondary Outcome: Stair Climbing Test (ST)
Description: Ascend and descend 8 steps with a step hight of 16 cm as fast as they could without running. Few seconds (best) - many seconds (worse)
Time Frame: 5 months and 12 months
Measure: Mean (95% Confidence Interval); unit: seconds
Groups:
- Walking Skill Training Group: 12 sessions of participation in the supervised walking skill training program
- Control Group: No sessions of participation in the walking skill training program
Arm/Group | Walking Skill Training Group | Control Group
Number analyzed (Participants) | 35 | 33
seconds
  ST at 5 months | 11 [10 to 11] | 12 [11 to 13]
  ST at 12 months | 10 [9 to 11] | 12 [11 to 13]

6. Secondary Outcome: ROM Extension
Description: Active range of motion (ROM) in hip extension test. Degrees is registered. 0 degrees indicates zero position of the hip, minus digrees indicates flexion contracture.
Time Frame: 5 months and 12 months
Measure: Mean (95% Confidence Interval); unit: degrees
Arm/Group | Walking Skill Training Group | Control Group
Number analyzed (Participants) | 35 | 33
degrees
  ROM extension at 5 months | 0 [-1 to 2] | -2 [-3 to -1]
  ROM extension at 12 months | 0 [-2 to 1] | -1 [-3 to 0]

7. Secondary Outcome: Index of Muscle Function (IMF)
Description: Tests of general mobility, muscle strength, balance/coordination, and endurance. 40 (worse) - 0 (best)
Time Frame: 5 months and 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Walking Skilll Training Group: 12 sessions of participation in the supervised walking skilll training program
Arm/Group | Walking Skilll Training Group | Control Group
Number analyzed (Participants) | 35 | 33
units on a scale
  IMF at 5 months | 8 [7 to 9] | 11 [9 to 12]
  IMF at 12 months | 7 [6 to 9] | 10 [8 to 11]

8. Secondary Outcome: Figure-of-eight Test
Description: Test of dynamic balance. Number of steps on and outside the line is registered. 0 (best)
Time Frame: 5 months and 12 months
Measure: Mean (95% Confidence Interval); unit: steps
Groups:
- Control Group: No session of participation in the walking skill training program
Arm/Group | Walking Skill Training Group | Control Group
Number analyzed (Participants) | 35 | 33
steps
  Figure-of-eight at 5 months | 7 [5 to 9] | 10 [8 to 12]
  Figure-of-eight at 12 months | 7 [5 to 8] | 8 [7 to 10]

ADVERSE EVENTS:
Time Frame: at 5 months (after the training program was completed) and at followup at 12 months
Description: No adverse events were registered
Arm/Group | Walking Skill Training Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/33
Other Adverse Events (participants affected / at risk) | 0/35 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No